CLINICAL TRIAL: NCT02478125
Title: A Pilot Study of Mobilization and Treatment of Disseminated Tumor Cells in Men With Metastatic Prostate Cancer
Brief Title: Pilot Study of Mobilization and Treatment of Disseminated Tumor Cells in Men With Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Prostate Cancer Foundation (Other); TaiGen Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J14177; IRB00054180 (Other: JHM IRB)
Record Dates: First submitted 2015-06-10; First posted 2015-06-23 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
Keywords: metastatic castrate resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- burixafor hydrobromide (Active Comparator): Four daily doses of burixafor hydrobromide alone
  Interventions: Drug: Burixafor Hydrobromide
- G-CSF (Active Comparator): G-CSF will be given as a daily subcutaneous (SC) injection beginning 4 days prior to Burixafor hydrobromide and continuing through the 4 days of Burixafor hydrobromide treatment
  Interventions: Drug: G-CSF
- Docetaxel (Experimental): Investigators will administer a single 75 mg/m2 IV dose of docetaxel. Twenty-one days later investigators will re-treat enrolled men with the optimal mobilization strategy + docetaxel IV.
  The second dose of docetaxel being given in combination with the optimal mobilization strategy will be chosen according to a standard 3+3 dose escalation schema, in which the dose of bruixafor +/- G-CSF will be held constant and the dose of docetaxel will escalate between three dose-levels: 1) docetaxel 30 mg/m2 IV, 2) docetaxel 60 mg/m2 IV, and 3) docetaxel 75 mg/m2
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Burixafor Hydrobromide — Investigators will determine the kinetics of PCa cell release into the blood with four daily dosages of Burixafor hydrobromide alone or in combination with G-CSF
  Arms: burixafor hydrobromide
Drug: Docetaxel — Investigators will administer a single 75 mg/m2 IV dose of docetaxel. Twenty-one days later investigators will re-treat enrolled men with the optimal mobilization strategy + docetaxel IV. The second dose of docetaxel being given in combination with the optimal mobilization strategy will be chosen according to a standard 3+3 dose escalation schema, in which the dose of bruixafor +/- G-CSF will be held constant and the dose of docetaxel will escalate between three dose-levels: 1) docetaxel 30 mg/m2 IV, 2) docetaxel 60 mg/m2 IV, and 3) docetaxel 75 mg/m2
  Arms: Docetaxel
Drug: G-CSF — G-CSF will be given as a daily subcutaneous (SC) injection beginning 4 days prior to Burixafor hydrobromide and continuing through the 4 days of Burixafor hydrobromide treatment
  Other Names: granulocyte-colony stimulating factor
  Arms: G-CSF

SUMMARY:
Hypothesis: Treatment with Burixafor hydrobromide will effectively mobilize metastatic prostate cancer (PCa) cells (i.e. disseminated tumor cells; DTCs) into the blood from the bone marrow. It has been demonstrated that prostate cancer cells have been mobilized out of the bone marrow of mice utilizing an anti-CXCR4 strategy; making them more susceptible to chemotherapy.

DETAILED DESCRIPTION:
This is an open label, multiple site, pilot study. Hypothesis: Treatment with Burixafor hydrobromide will effectively mobilize metastatic prostate cancer (PCa) cells (i.e. disseminated tumor cells; DTCs) into the blood from the bone marrow. In preclinical models, these bone marrow niche engaged cells are more resistant to therapy as compared to soft tissue sites.

It has been demonstrated that prostate cancer cells have been mobilized out of the bone marrow of mice utilizing an anti-CXCR4 strategy; making them more susceptible to chemotherapy. Currently, the anti-CXCR4 agent plerixafor is FDA approved to be given for up to 4 consecutive days in order to mobilize hematopoietic stem cells (HSCs).

Burixafor hydrobromide is a potent anti-CXCR4 agent that is in clinical trials. Burixafor hydrobromide, alone or in combination with G-CSF, is currently in Phase II testing for use as a hematopoetic stem cell (HSC) mobilization agent. When Burixafor hydrobromide is given intravenously (IV) alone at a dose of 3.14 mg/kg it has been shown to result in a 7.8 fold mean increase in peripheral blood CD34+ (a HSC marker) cells 6-hours post-infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Have signed an informed consent document indicating that the subject understands the purpose of and procedures required for the study and are willing to participate in the study
2. Be willing/able to adhere to the prohibitions and restrictions specified in this protocol
3. Male aged 18 years and above
4. Eastern cooperative group (ECOG) performance status ≤2
5. Documented histologically confirmed adenocarcinoma of the prostate
6. Metastatic prostate cancer to the bone as documented by positive bone scan imaging
7. Patient must be eligible for chemotherapy with docetaxel
8. Patient must have evidence of castrate resistant prostate cancer as evidenced by a confirmed rising PSA (per Prostate Cancer Working Group 2 [PCWG2] criteria) and a castrate serum testosterone level (i.e. ≤ 50 mg/dL).

Exclusion Criteria:

1. Have known allergies, hypersensitivity, or intolerance to docetaxel or dexamethasone or their excipients
2. Prior pelvic radiation (e.g. external beam, brachytherapy, etc) that, in the opinion of the investigator, may lead to decreased bone marrow cellularity in a marrow sample obtained from a pelvic bone marrow biopsy
3. Ongoing systemic therapy (other than a GnRH agonist/antagonist) for prostate cancer including, but not limited to:

   1. CYP-17 inhibitors (e.g. ketoconazole, abiraterone)
   2. Antiandrogens (e.g. bicalutamide, nilutamide)
   3. Second generation antiandrogens (e.g. enzalutamide)
   4. Immunotherapy (e.g. sipuleucel-T, ipilimumab)
   5. Chemotherapy (e.g. docetaxel, cabazitaxel)
4. Prior radiopharmaceutical therapy (e.g. radium-223, strontium-89, samarium-153, etc) within the past year
5. Have any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements
6. Active infection or other medical condition that would make corticosteroids (i.e. dexamethasone) use contraindicated
7. Uncontrolled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg) Patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment
8. Severe hepatic impairment (Child-Pugh Class C)
9. History of pituitary or adrenal dysfunction (note: the use of daily steroids does not exclude someone from participating in this study)
10. Have poorly controlled diabetes (HgB A1C ≥ 8%)
11. Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Mobilization of DTCs from bone marrow | 2 years
  Measure the number of CTCs in the peripheral blood.

SECONDARY OUTCOMES:
Kinetics of disseminated tumor cell mobilization by quantifying the number of circulating tumor cells per milliliter of blood over time | 2 years
  This will be reported as number of tumor cells/mL at multiple time points following infusion of Burixafor hydrobromide with and without G-CSF.
Kinetics of hematopoietic stem cell (HSC) mobilization by quantifying the number of circulating HSCs per milliliter of blood over time | 2 years
  This will be reported as number of HSC/mL at multiple time points following infusion of Burixafor hydrobromide with and without G-CSF.
PSA response to treatment with Burixafor hydrobromide alone and Burixafor hydrobromide and docetaxel | 2 years
Safety of Burixafor hydrobromide +/- GCSF +/- docetaxel | 2 years
  Safety will be evaluated by the incidence, severity, duration, causality, seriousness, and type(s) of adverse events
Exploratory biomarker Assessment on CTCs/DTCs | 2 years
  Examples of these may include, but are not limited to: assessment of cell cycle kinetics, apoptosis, PTEN status, MYC alterations, whole genome, whole exome, and transcriptome analysis

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Pienta, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States